CLINICAL TRIAL: NCT01127425
Title: Length of Hospital Stay, Nursing Hours and Recovery After Laparoscopic Versus Open Colon Resection Without Fast Track
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to reorganisation in the hospital structure
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Doctor Britta Kaltoft, Gentofte Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA-20060067
Record Dates: First submitted 2010-02-17; First posted 2010-05-20 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2006-06

CONDITIONS: Sigmoid Neoplasms
Keywords: nursing hours; length of hospital stay; reconvalescence; colorectal surgery; laparoscopic; sigmoid neoplasms
MeSH Terms: conditions — Sigmoid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Intervention: Surgery: laparoscopic sigmoid resection without fast track postoperative care
  Interventions: Procedure: laparoscopic sigmoid resection
- 2 (Active Comparator): Intervention: Surgery: conventional (open) sigmoid resection without fast track postoperative care
  Interventions: Procedure: laparoscopic colonic resection

INTERVENTIONS:
Procedure: laparoscopic colonic resection — Conventional surgery compared to laparoscopic sigmoid resection
  Arms: 2
Procedure: laparoscopic sigmoid resection — sigmoid resection by laparoscopic surgery
  Arms: 1

SUMMARY:
A blinded randomized trial. Length of hospital stay, nursing hours and recovery after laparoscopic versus open colonic resection without fast track.

DETAILED DESCRIPTION:
CONTEXT: Our preliminary experience (unpublished) indicate that less nursing hours are needed after laparoscopic colon resection without fast track. Length of hospital stay and recovery seems to be reduced as well.

OBJEKTIVE: To compare laparoscopic and open colonic resection concerning nursing hours, length of hospital stay and recovery.

DESIGN, SETTING AND PATIENTS: triple blinded study (Patient, nursing staff and data collector) including 2 x 12 patients needing sigmoid resection due to cancer. Nursing hours, length of hospital stay and recovery (postoperative pain, questionnaire, actigraph ect.)

ELIGIBILITY:
Inclusion Criteria:

* sigmoid resection without stoma
* sigmoid neoplasms localized 20 cm from anus
* age 40-90

Exclusion Criteria:

* conversion from laparoscopic to open surgery
* stoma
* severe postoperative complications (anastomosis leak, intraabdominal abscess, reoperation, stay at intensive care unit, heart attack, pulmonary embolism)
* no informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
primary: Length of stay | 1 year

SECONDARY OUTCOMES:
secondary: Nursing hours, pain and recovery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Britta Kaltoft, doctor, Principal Investigator — University of Gentofte
Locations (1):
- University Hospital of Gentofte, gastroenterologic surgery, Hellerup, Denmark